CLINICAL TRIAL: NCT02956603
Title: Studying Electromyographic Activity in Patients With Upper Limb Amputations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Paul Cederna, Robert Oneal Professor and Chief of Plastic Surgery; Professor, Biomedical Engineering, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00088547; N66001-16-1-4006 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Amputation, Traumatic
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neuroma Graft (Experimental): In this arm, participants have already had partial muscle grafts placed on the amputated nerves to control neuroma growth. The investigators will place small electrodes percutaneously into the muscle grafts to record EMG signals and electrically stimulate the implanted nerves.
  Interventions: Other: Fine wire EMG electrodes
- Prosthetic Control Graft (Experimental): In this arm, participants will have an initial surgery to place partial muscle grafts on the amputated nerves. After a healing period, the investigators will place small electrodes percutaneously into the muscle grafts to record EMG signals and electrically stimulate the implanted nerves.
  Interventions: Other: Fine wire EMG electrodes
- Able Bodied (Experimental): The investigators will place small electrodes percutaneously into intact muscles in the arm to record EMG signals and electrically stimulate the intact nerves nearby.
  Interventions: Other: Fine wire EMG electrodes

INTERVENTIONS:
Other: Fine wire EMG electrodes — Electrodes placed either in partial muscle grafts or in intact muscle to record and stimulate

SUMMARY:
The primary purpose of this study is to determine the extent to which the Regenerative Peripheral Nerve Interface ( i.e. reinnervation of partial muscle grafts by residual peripheral nerves) enables both the generation of high-performance motor control signals for prosthetic limbs, and the input of sensory percepts by electrical stimulation.

ELIGIBILITY:
Inclusion criteria:

* For the prosthetic control graft arm:

  * Must have previously undergone upper limb amputation
  * Must be otherwise healthy (e.g. no severe pain syndromes or untreated mental health disorders)
  * Must be American Society of Anesthesiologists (ASA) Class I (low surgical risk)
  * Must have sufficient soft tissue quality to support performance of the operative procedures
  * Must have NOT previously received the partial muscle graft surgery
* For the neuroma graft arm:

  * Must have previously undergone upper limb amputation
  * Must be otherwise healthy (e.g. no severe pain syndromes or untreated mental health disorders)
  * Must have previously received the partial muscle graft surgery
* For the able-bodied arm:

  * Must have NOT undergone upper limb amputation
  * Must be in good health

Exclusion criteria:

* For the prosthetic control graft arm:

  * Participants sustaining severe crushing or avulsion injuries with substantial superficial and deep scarring, may not be appropriate candidates for inclusion in the study
* For the able-bodied arm:

  * Participants with a history of nerve pain may not be appropriate candidates for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-06 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Amplitude of EMG signal | <4 hours
Number of separate sensory percepts evoked | <4 hours

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared